CLINICAL TRIAL: NCT06219616
Title: Prediction of BK Virus Infection by Flow Cytometric Analysis of BK Virus-specific T Cell Responses in Kidney Transplant Recipients
Brief Title: Prediction of BK Virus Reactivation in Kidney Transplant Recipient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Suwasin Udomkarnjananun, Assistant Professor, King Chulalongkorn Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: BKV-KCMH
Record Dates: First submitted 2024-01-04; First posted 2024-01-23 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-03

CONDITIONS: Kidney Transplant Infection; BK Virus Infection; BK Virus Nephropathy

STUDY DESIGN:
Intervention Model Description: Every kidney transplant recipient will be tested for BKV-specific immune response after transplantation to identify the potential immune predicting tool for developing BKV reactivation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BKV immune monitoring (Other): 1. In this prospective cohort, the included kidney transplant recipients will receive regular post-transplantation care, including routine therapeutic drug monitoring of tacrolimus and screening for BK viremia. No extra medications beyond the standard of care will be given to the patients in this study.
  2. Whole blood will be drawn from kidney transplant recipients on day 30, day 180, and at the time of BK viremia. PBMCs will be separated and incubated with BK viral peptides.
  3. PBMCs will be stained for surface marker of activated T cells and intracellular cytokines 4. Phenotypic features of T cells will be analyzed under flow cytometry and correlated with the occurrence of BKV infection and immunosuppressive medications.
  Interventions: Diagnostic Test: BKV immune monitoring

INTERVENTIONS:
Diagnostic Test: BKV immune monitoring — Blood will be drawn and investigated for BKV-specific T cell response.

SUMMARY:
There has been no effective predicting tool to accurately predict BKV reactivation after kidney transplantation. The aim is to elucidate the use of flow cytometric analysis for both intracellular cytokines and surface activation markers for BKV-specific T cell response in kidney transplant recipients.

ELIGIBILITY:
Inclusion criteria:

1. New kidney transplantation cases (either living donor or deceased donor transplantation)
2. Age ≥ 18 years old
3. Agree to give a permission to blood sampling post-transplantation, and at the time of BK viremia.

Exclusion criteria:

1. Pregnant
2. Primary non-function of kidney allograft (i.e. kidney allograft never function).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
BKV-specific immune response | Day 30, Day 90 after transplantation before BK viremia
  - To examine the capability of flow cytometry in predicting post-kidney transplant BKV infection, by the analyses of intracellular cytokines (interleukine-2) and surface activation markers (CD25) of T cells

SECONDARY OUTCOMES:
Dynamic change of BKV-specific immune response | Day 30, Day 90 after transplantation, irrespective ly to BK viremia
  To examine the chonological change of BKV-specific immune response after transplantation, by the analyses of intracellular cytokines (interleukine-2) and surface activation markers (CD25) of T cells.
BKV-specific immune response and immunosuppression regimen | Day 30, Day 90 after transplantation, in correlation to immunosuppressive medications
  To examine the association between immunosuppressive regimen (tacrolimus, cyclosporine A, mycophenolate) and BKV-specific immune response after transplantation, by the analyses of intracellular cytokines (interleukine-2) and surface activation markers (CD25) of T cells.

CONTACTS AND LOCATIONS:
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided